CLINICAL TRIAL: NCT05637450
Title: Blue Whiting Protein Hydrolysates and Sarcopenia Outcomes in Older Adults Residing in Residential Care Facilities (SARCO_CARE)
Brief Title: Fish Protein Supplementation and Sarcopenia Outcomes in Carehomes
Acronym: SARCO_CARE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Ulster (Other)
Collaborators: University of Limerick (Other); Bio-Marine Ingredients Ireland (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 22/NI/0108
Record Dates: First submitted 2022-11-21; First posted 2022-12-05 (Actual); Last update posted 2022-12-05 (Actual); Status verified 2022-12

CONDITIONS: Sarcopenia
Keywords: Sarcopenia; Fish protein; Fish hydrolysates; Protein supplementation; Older adults; Community; Muscle strength
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Intervention Model Description: Double-blind randomised control trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants are assigned to intervention groups by chance
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fish protein supplement (Experimental): Blue Whiting Protein Hydrolysate
  Interventions: Dietary Supplement: Blue Whiting Protein Hydrolysate
- Placebo (Placebo Comparator): Isocalorific Maltodextrin Citrus Flavoured Powder
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Blue Whiting Protein Hydrolysate — 25g Blue Whiting Protein Hydrolysates mixed with an everyday food / drink product daily for 6 weeks
  Arms: Fish protein supplement
Dietary Supplement: Placebo — Isocalorific maltodextrin citrus flavoured powder mixed with an everyday food / drink product for 6 weeks
  Arms: Placebo

SUMMARY:
The proposed study aims to investigate the effect of consuming 12.5g (twice daily) Blue Whiting Protein Hydrolysates (BWPH) daily for 6 weeks on whole body lean mass tissue and measures of muscle strength and functionality in older adults residing in residential care facilities.

DETAILED DESCRIPTION:
Sarcopenia is a progressive and generalised skeletal muscle disorder involving the accelerated loss of muscle mass and function that is associated with increase adverse outcomes including falls, functional decline, frailty and mortality. Diet, specifically protein has been proposed to have a role in the prevention and treatment of muscle loss in the older adult population nevertheless there is paucity of research on the effect of protein supplementation on lean body mass and other clinical outcomes in older adults, and especially those in residential care where the prevalence of muscle loss and weakness is reported to be high This 2-arm parallel, double-blind, randomised, controlled dietary supplement human intervention study aims to investigate the effect of consuming 12.5g (twice daily) Blue Whiting Protein Hydrolysates daily for 6 weeks on whole body lean mass tissue and measures of muscle strength and functionality in free living community dwelling older adults. A total of 184 participants (92 per group) is required based on a previous study by Norton et al (2015) Participants will be stratified by age, gender and BMI and randomly allocated to consume two sachets of either the BWPH powder daily (12.5g at lunch and dinner (Total 25g)), (mixed with an everyday food / drink product (provided by Ulster University) or an isocalorific maltodextrin citrus flavoured powder (Control) (mixed with an everyday food / drink product).

Assessments to be undertaken pre and post intervention include; body composition including lean mass tissue by Tanita body composition monitor, hand grip strength, a 'timed get up and go' test, chair stand test, blood pressure measurements, a habitual dietary intake questionnaire, quality of life questionnaire, SARC-F (screening tool for sarcopenia) and an MNA questionnaire (mini nutritional assessment). A trained phlebotomist will obtain a 40ml max blood sample from each participant pre and post intervention. Blood samples will be used to measure markers associated with sarcopenia (serum 25(OH)D, pro inflammatory cytokine profile, full lipid profiles and kidney and liver profiles).

All researchers taking physical measurements will be trained in the correct procedure and will follow a standardised protocol whilst taking all measurements. All physical measurements will be taken with the participant wearing light clothing (without footwear). Measurements will be taken pre- and post-intervention unless otherwise stated. All measurements for each participant will be recorded on a single data collection sheet.

Height and weight will be measured to determine BMI (kg/m2). Standing height (m) will be measured (pre-intervention only) to the nearest 0.5cm using a calibrated stadiometer (SECA, Model 220, Germany). Body weight (kg) will be recorded without footwear or heavy clothing and measured to the nearest 0.1kg using portable scales (Seca; Brosch Direct Ltd, Peterborough, UK).

A Tanita body composition monitor will use bioelectrical impedance analysis to estimate body composition in all participants, except in those with pacemakers because of the electrical current used.

Blood pressure will be measured using an Omron 705CP electronic blood pressure monitor (Medisave, Dorset, UK). A reading will be taken from both arms of each participant, and the arm with the highest reading for each individual will subsequently be used as the reference arm. A mean of two blood pressure readings (taken at least 10 minutes apart while the subject is seated and at-rest) will be taken from the same reference arm at all appointments. A third measurement will be taken if the first two measurements deviate by more than 10%.

Hand grip dynamometry will be used to assess grip strength (kg) as a measure of upper body muscle function and will be measured on the non-dominant side three times. In a standing position, with arms at their side (not touching the body and keeping elbows slightly bent), the participant will be asked to hold the device and grip as tightly as possible whilst raising their arm out to the side, taking care to only squeeze once for each measurement. There will be a 10-20 second rest between measurements.

A timed up & go test will be conducted to test basic mobility (Podsiadlo & Richardson, 1991). A 3 metre distance will be identified and the participant will be asked to stand up from a chair, walk at a normal pace to the line on the floor which is 3 metres from the chair, turn, walk back to the chair at normal pace and sit down again. The time taken to do this will be recorded. A trained researcher will explain the exact procedure to the participant.

A chair stand test will be conducted to assess functional fitness. Participants will be instructed to perform five rises with arms crossed resting hands on their shoulders, moving from a seated position to a stand position. The amount of time spent to perform the test will be reported.

The planned statistical analysis will be conducted using the Statistical Package for the Social Sciences (SPSS) for Windows version 24.0 (SPSS Inc, Chicago, IL, USA). Intention to treat analysis will be used. Descriptive statistics will be used to present characteristics pre- and post- intervention. Comparisons will be made (ANCOVA) between the intervention group and control group over time.

ELIGIBILITY:
Inclusion Criteria:

* Individuals residing in a residential care facility
* Willing to participate in the study
* Without major cognitive impairment
* Not regularly taking protein supplements
* Not at end-of-life stage

Exclusion Criteria:

* At end-of-life stage.
* Major cognitive impairment
* Exclusively receiving enteral or parenteral nutrition
* Food allergy or intolerance that would prevent consumption of the study supplement (e.g. fish)
* Currently taking any protein supplement

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 184 (Estimated)
Dates: Start 2023-07-01 (Estimated); Primary Completion 2023-08-31 (Estimated); Study Completion 2023-08-31 (Estimated)

PRIMARY OUTCOMES:
Lean mass | Change over 6 weeks
  Assessed via Tanita body composition monitor

SECONDARY OUTCOMES:
Muscle strength | Change over 6 weeks
  Measured via hand grip dynamometry
Muscle functionality | Change over 6 weeks
  Measured via hand grip dynamometry
Mobility | Change over 6 weeks
  Assessed through timed get up and go test (time to walk 3 metres)
Mobility | Change over 6 weeks
  Assessed through chair stand test

OTHER OUTCOMES:
General clinical chemistry | Change over 6 weeks
  Full lipid profile (Total, HDL & triacylglycerols) measured photometrically on an automatic analyser. LDL will be calculated by the Friedewald formula
General clinical chemistry | Change over 6 weeks
  Vitamin B status
General clinical chemistry | Change over 6 weeks
  Vitamin D status
General clinical chemistry | Change over 6 weeks
  Pro inflammatory markers (Human panel 1) measured on Meso Scale Discovery

IPD SHARING:
Plan to Share IPD: No
Company funded research